CLINICAL TRIAL: NCT07257679
Title: The Effects of 'Gentle Touch' in the Management of Lymphedema in Women Treated for Breast Cancer: A Preliminary Single-blind, Parallel-group Randomized Controlled Trial.
Brief Title: Gentle Touch for Post-Mastectomy Lymphedema
Acronym: GT-BCRL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Comitato A.N.D.O.S. di Roma odv. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 387/SL/25
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Lymphedema, Breast Cancer
Keywords: Lymphedema; Breast Cancer; DLM; Gentle touch
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentle Touch (GT) Lymphatic Drainage + Usual Care (Experimental): Participants in this arm will receive the Gentle Touch (GT) lymphatic drainage technique, which is based on the ANDOS manual technique, in addition to their existing rehabilitation pathway. The GT is a tactile stimulus applied to the skin aimed at promoting relaxation, improving pain, sleep management, and therapeutic participation. The treatment involves 10 sessions administered with a bi-weekly frequency.
  Interventions: Other: Gentle Touch (GT) Lymphatic Drainage (ANDOS technique)
- Passive Mobilization and Active-Assisted Exercises + Usual Care (Active Comparator): Participants in this arm will receive 10 sessions of passive mobilization and active-assisted exercises for the upper limb. This is provided in addition to the existing rehabilitation program. The sessions will be carried out with the same frequency (bi-weekly) as the experimental group.
  Interventions: Other: Passive Mobilization and Active-Assisted Exercises for the Upper Limb

INTERVENTIONS:
Other: Gentle Touch (GT) Lymphatic Drainage (ANDOS technique) — This intervention involves the application of a specific tactile stimulus (Gentle Touch) to the skin. This stimulus is designed to promote relaxation, alleviate social isolation and stress, and provide emotional support. The goal is to stimulate fluid movement in the skin, increasing lymphatic flow, attenuating fibrosis, and reducing pain. This approach (GT-based ANDOS technique) is added to the participant's existing rehabilitation program. The intervention is administered by a specifically trained physiotherapist. Dosage: 10 sessions. Frequency: Bi-weekly.
  Arms: Gentle Touch (GT) Lymphatic Drainage + Usual Care
Other: Passive Mobilization and Active-Assisted Exercises for the Upper Limb — This intervention consists of passive mobilization and active-assisted exercises for the affected upper limb. This intervention is given in addition to the participant's existing rehabilitation program. This is the control intervention to which the experimental GT approach is compared. It is administered by a specifically trained physiotherapist. Dosage: 10 sessions. Frequency: Bi-weekly (same as the experimental group).
  Arms: Passive Mobilization and Active-Assisted Exercises + Usual Care

SUMMARY:
This is a single-blind, parallel-group Randomized Controlled Trial (RCT) comparing the efficacy of a specialized manual technique, Gentle Touch (GT), versus a control intervention, both added to the usual rehabilitative care. The study investigates 36 women aged 30 to 75 with Breast Cancer-Related Lymphedema (BCRL). The primary objective is to evaluate the reduction of lymphedema volume in the upper limb. Secondary objectives include assessing the improvement in patients' quality of life and the potential reduction in care burden and costs. The treatment protocol involves 10 bi-weekly sessions over 5 weeks.

DETAILED DESCRIPTION:
Breast cancer (BC) treatment often leads to lymphedema, a condition affecting up to 40% of survivors and negatively impacting their quality of life due to swelling, pain, and functional limitations. Manual Lymphatic Drainage (MLD) is a proven treatment method. This study focuses on the Gentle Touch (GT) approach, a specific tactile stimulus applied to the skin intended to promote emotional support, relaxation, and stress alleviation.

The Primary Objective is to evaluate the efficacy of the Gentle Touch-based MLD in reducing the volume of upper limb lymphedema in women who have undergone surgery for BC.

The Secondary Objectives are to evaluate whether the GT approach can improve the quality of life of the treated women, including emotional, psychological, and social aspects and reduce the care burden and costs compared to the control group, potentially by reducing the number of treatments required compared to conventional approaches.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Women.
* Age: Between 30 and 75 years old
* Surgical History: Women who have undergone surgery for breast cancer (BC). This includes being subjected to one of the following interventions: Axillary dissection with removal of all 3 lymph node levels; Axillary dissection with removal of only one lymph node level; Removal of the sentinel lymph node only.
* Clinical Lymphedema: Clinically evaluated lymphedema symptoms, defined as a circumference difference of greater than 20mm between the two arms

Exclusion Criteria:

* Concurrent Diseases: Concomitant diseases that may interfere with the study.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change of Upper Limb Lymphedema Volume | Baseline (T0), 5 weeks (T1), and 2-month follow-up (T2)
  The volume of lymphedema will be measured volumetrically, comparing the difference in volume of the affected limb relative to the contralateral limb.

SECONDARY OUTCOMES:
Change in Lymphedema-Specific Quality of Life (LYMQOL) | Baseline (T0), 5 weeks (T1), and 2-month follow-up (T2)
  Measured using the Lymphoedema Quality of Life Questionnaire (LYMQOL) score. Scores on the LYMQOL range from 1 to 4 for each item, with a total score ranging from 21 to 84; higher scores indicate a worse quality of life.
Change in Upper Limb Function and Disability (DASH) | Baseline (T0), 5 weeks (T1), and 2-month follow-up (T2)
  Measured using the total score of the Disability of the Arm Shoulder and Hand Questionnaire (DASH). DASH scores range from 0 to 100, with higher scores indicating greater disability and thus worse upper limb function and quality of life.
Change in General Health (SF-36) | Baseline (T0), 5 weeks (T1), and 2-month follow-up (T2)
  Measured using the scores of the SF-36 Questionnaire general health. SF-36 scores range from 0 to 100; higher scores indicate better health status (i.e. better perceived quality of life / functioning)
Change in Well-being (PROMIS-29) | Baseline (T0), 5 weeks (T1), and 2-month follow-up (T2)
  Measured using the scores of the PROMIS-29 Questionnaire, to assess general physical and mental health status. PROMIS-29 provides scores for seven health domains. For each domain, raw scores range from 4 to 20. Higher scores indicate better outcomes for physical function and social participation, and worse outcomes for pain, fatigue, depression, anxiety, and sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Santa Lucia Foundation IRCCS, Roma, RM
  - Santa Lucia Foundation, Scientific Institute for Research and Health Care, Roma, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loibl S, Andre F, Bachelot T, Barrios CH, Bergh J, Burstein HJ, Cardoso MJ, Carey LA, Dawood S, Del Mastro L, Denkert C, Fallenberg EM, Francis PA, Gamal-Eldin H, Gelmon K, Geyer CE, Gnant M, Guarneri V, Gupta S, Kim SB, Krug D, Martin M, Meattini I, Morrow M, Janni W, Paluch-Shimon S, Partridge A, Poortmans P, Pusztai L, Regan MM, Sparano J, Spanic T, Swain S, Tjulandin S, Toi M, Trapani D, Tutt A, Xu B, Curigliano G, Harbeck N; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Early breast cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2024 Feb;35(2):159-182. doi: 10.1016/j.annonc.2023.11.016. Epub 2023 Dec 13. No abstract available. PMID 38101773
- [Background] Fu MR, Ridner SH, Hu SH, Stewart BR, Cormier JN, Armer JM. Psychosocial impact of lymphedema: a systematic review of literature from 2004 to 2011. Psychooncology. 2013 Jul;22(7):1466-84. doi: 10.1002/pon.3201. Epub 2012 Oct 9. PMID 23044512
- [Background] Thompson B, Gaitatzis K, Janse de Jonge X, Blackwell R, Koelmeyer LA. Manual lymphatic drainage treatment for lymphedema: a systematic review of the literature. J Cancer Surviv. 2021 Apr;15(2):244-258. doi: 10.1007/s11764-020-00928-1. Epub 2020 Aug 15. PMID 32803533
- [Background] Sezer Efe Y, Erdem E, Caner N, Gunes T. The effect of gentle human touch on pain, comfort and physiological parameters in preterm infants during heel lancing. Complement Ther Clin Pract. 2022 Aug;48:101622. doi: 10.1016/j.ctcp.2022.101622. Epub 2022 Jun 22. PMID 35759976